CLINICAL TRIAL: NCT00943826
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase III Trial of Bevacizumab, Temozolomide and Radiotherapy, Followed by Bevacizumab and Temozolomide Versus Placebo, Temozolomide and Radiotherapy Followed by Placebo and Temozolomide in Patients With Newly Diagnosed Glioblastoma
Brief Title: A Study of Bevacizumab (Avastin®) in Combination With Temozolomide and Radiotherapy in Participants With Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BO21990; 2008-006146-26 (EudraCT Number)
Record Dates: First submitted 2009-07-17; First posted 2009-07-22 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-08

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; Temozolomide; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Bevacizumab + RT + Temozolomide (Experimental): In the Concurrent Phase participants will receive radiotherapy (RT) in daily fractions of 2 Gy to be given 5 days per week for 6 weeks and temozolomide 75 mg/m^2 daily from the first day to the last day of radiotherapy (it may continue for a maximum of 49 days in case of delay to the end of radiation therapy) and bevacizumab 10 mg/kg IV every 2 weeks for 6 weeks. There will be a 4 week treatment break. Participants will then enter the Maintenance Phase where they receive six 28-day cycle of bevacizumab 10 mg/kg IV q2w and temozolomide 150 to 200 mg/m^2 daily in the first 5 days of each cycle. The participants will then enter the Monotherapy Phase where they will receive bevacizumab 15 mg/kg IV q3w until disease progression/unacceptable toxicity.
  Interventions: Drug: Bevacizumab; Drug: Temozolomide; Radiation: Radiation therapy
- Placebo + RT + Temozolomide (Placebo Comparator): In the Concurrent Phase participants will receive radiotherapy in daily fractions of 2 Gy to be given 5 days per week for 6 weeks and temozolomide 75 mg/m^2 daily from the first day to the last day of radiotherapy (it may continue for a maximum of 49 days in case of delay to the end of radiation therapy) and placebo IV every 2 weeks for 6 weeks. There will be a 4 week treatment break. Participants will then enter the Maintenance Phase where they will receive six 28-day cycle of placebo IV q2w and temozolomide 150 to 200 mg/m^2 daily in the first 5 days of each cycle. The participants will then enter the Monotherapy Phase where they will receive placebo IV q3w until disease progression/unacceptable toxicity.
  Interventions: Drug: Temozolomide; Radiation: Radiation therapy; Drug: Placebo

INTERVENTIONS:
Drug: Bevacizumab — 10 mg/kg intravenously q2w in the Concurrent and Maintenance Phases. 15 mg/kg intravenously q3w in the Monotherapy Phase.
  Other Names: Avastin
  Arms: Bevacizumab + RT + Temozolomide
Drug: Temozolomide — 75 mg/m^2 once daily for 6 weeks, followed by 150-200 mg/m^2 once daily on days 1-5 of six 4 week cycles.
Radiation: Radiation therapy — 30 fractions of 2 Gy delivered on days 1-5 per week for 6 weeks.
Drug: Placebo — Intravenously q2w in the Concurrent and Maintenance Phases and q3w in the Monotherapy Phase.
  Arms: Placebo + RT + Temozolomide

SUMMARY:
This 2 arm study investigated the efficacy and safety of the addition of bevacizumab to the current standard of care (multimodality therapy of concurrent radiotherapy plus temozolomide followed by adjuvant temozolomide) as compared to the current standard of care alone. Participants were randomly assigned to either the bevacizumab (10 milligrams per kilogram (mg/kg) intravenously [IV] once every 2 week [q2w]) or the placebo arm, in combination with radiation therapy (total dose 60 Gray [Gy], administered as 2 Gy fractions, 5 days/week) plus temozolomide (75 milligrams per meter squared [mg/m^2] oral administration [po] daily) for 6 weeks. After a 4 week treatment break, participants continued to receive bevacizumab (10 mg/kg IV q2w) or placebo, plus temozolomide (150-200 mg/m^2 po daily on days 1-5 of each 4 week cycle) for 6 cycles of maintenance treatment or until disease progression or unacceptable toxicity, whichever occured first. Following the maintenance phase, bevacizumab (15 mg/kg iv every 3 weeks [q3w]) or placebo monotherapy continued. The time on study treatment was until disease progression.

ELIGIBILITY:
Key Inclusion Criteria:

* newly diagnosed glioblastoma
* World Health Organization (WHO) performance status less than or equal to (<=2)
* stable or decreasing corticosteroid dose within 5 days prior to randomization

Key Exclusion Criteria:

* evidence of recent hemorrhage on postoperative magnetic resonance imaging (MRI) of brain
* any prior chemotherapy or immunotherapy for glioblastomas and low grade astrocytomas
* any prior radiotherapy to brain
* clinically significant cardiovascular disease
* history of greater than or equal to (>=) grade 2 hemoptysis within 1 month prior to randomization
* previous centralized screening for Methylguanine-DNA methyltransferase (MGMT) status for enrollment into a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 921 (Actual)
Dates: Start 2009-06-29 (Actual); Primary Completion 2013-02-28 (Actual); Study Completion 2015-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (133):
- United States (9):
  - University of Alabama At Birmingham; Neuro-Oncology, Birmingham, Alabama
  - UCLA, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Oncology-Evanston Nthwest Healthcare Kellogg Cancer Care Ctr, Evanston, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - Hatton Research Institutes, Cincinnati, Ohio
  - Sarah Cannon Cancer Center and Research Institute, Nashville, Tennessee
  - University of Virgina, Charlottesville, Virginia
- Australia (7):
  - Prince of Wales Hospital; Department of Medical Oncology, Randwick, New South Wales
  - North Shore Private Hospital; Northern Specialist Centre, St Leonards, New South Wales
  - Royal North Shore Hospital; Department of Medical Oncology, St Leonards, New South Wales
  - Princess AleXandra Hospital; Department of Medical Oncology, Woolloongabba, Queensland
  - Calvary North Adelaide; North Adeliade Oncology Centre, North Adelaide, South Australia
  - Royal Melbourne Hospital; Hematology and Medical Oncology, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Belgium (6):
  - Clin Univ de Bxl Hôpital Erasme, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Antwerpen, Edegem
  - AZ Sint Lucas (Sint Lucas), Ghent
  - CHU Sart-Tilman, Liège
  - AZ Delta (Campus Wilgenstraat), Roeselare
- Canada (14):
  - Tom Baker Cancer Centre-Calgary, Calgary, Alberta
  - Cross Cancer Institute ; Dept of Medical Oncology, Edmonton, Alberta
  - BC Cancer Agency, Vancouver Clinic; Dept. of Medical Oncology, Vancouver, British Columbia
  - CancerCare Manitoba; Neuro-Oncology, Winnipeg, Manitoba
  - Hamilton Health Sciences - Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario; Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre; Neuro-Oncology, Ottawa, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital; Pencer Brain Tumour Centre, 18-727, Toronto, Ontario
  - Hopital Notre-Dame, Montreal, Quebec
  - McGill University; Montreal Neurological Institute; Oncology, Montreal, Quebec
  - Chuq - Hopital Hotel Dieu de Quebec, Québec, Quebec
  - Saskatoon Cancer Centre; Uni of Saskatoon Campus, Saskatoon, Saskatchewan
- Denmark (3):
  - Aalborg Universitetshospital, Klinik Kirurgi-Kræft, Onkologisk afd., Aalborg
  - Righospitalet, Hæmatologisk Klinik, København Ø
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense
- France (11):
  - Hopital Avicenne; Rhumatologie, Bobigny
  - Hopital Saint Andre; Département de Radiothérapie Et D'Oncologie Médicale, Bordeaux
  - Institut Bergonie; Gastro Enterologie Oncologie, Bordeaux
  - Hopital neurologique Pierre Wertheimer - CHU Lyon; Neurologie, Bron
  - Centre Jean Perrin; Hopital De Jour, Clermont-Ferrand
  - Hopital Beaujon; Oncologie, Clichy
  - Centre Georges François Leclerc, Dijon
  - Hopital de La Timone - CHU de Marseille; Service de neuro-oncologie - Hôpital Adultes - 12ème étage, Marseille
  - Centre Val Aurelle Paul Lamarque; Medecine B3, Montpellier
  - Hôpital Central; Departement de Neuro-Oncologie, Nancy
  - Hopital Pitié Salpétrière - CHU; Service de neurologie 2 - Mazarin, Paris
- Germany (7):
  - Universitätsklinikum "Carl Gustav Carus"; Klinik und Poliklinik für Neurochirurgie, Dresden
  - Justus-Liebig-Universität Giessen; Neurochirurgische Klinik, Giessen
  - Universitatsklinikum Hamburg-Eppendorf; Klinik und Poliklinik fur Neurochirurgie, Hamburg
  - Universitatsklinikum Heidelberg; Abteilung Neuroonkologie, Heidelberg
  - Ärztehaus Velen, Ibbenbühren
  - Klinikum der Johannes Gutenberg Uni Mainz; Studienz. Neurologie, Klinik und Poliklinik Neurologie, Mainz
  - Uni Klinikum München - Großhardern; Med. Klinik U. Poliklinik III - Abt. Onkologie u. Hämatologie, München
- Greece (3):
  - Univ General Hosp Heraklion; Medical Oncology, Heraklion
  - University Hospital of Larissa; Oncology, Larissa
  - Papageorgiou General Hospital; Medical Oncology, Thessaloniki
- Hong Kong (3):
  - Dr Stephen Yau; Clinical oncology, Hong Kong
  - Hong Kong Sanatorium & Hospital; Comprehensive Oncology Centre, Hong Kong
  - Queen Mary Hospital; Microbiology Dept., Hong Kong
- Hungary (3):
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktató Kórház; Neurosurgery, Miskolc
  - Pécsi Tudományegyetem Áok; Onkoterapias Intezet, Pécs
- Israel (4):
  - Rambam Medical Center; Oncology, Haifa
  - Hadassah Hebrew University Hospital; Leslie and Michael Gaffin Center for Neuro-Oncology, Jerusalem
  - Rabin MC; Davidof Center - Oncology Institute, Petah Tikva
  - Chaim Sheba MC; Pediatric Hematology Oncology, Tel Litwinsky
- Italy (6):
  - Ausl Di Bologna-Ospedale Bellaria;U.O. Oncologia Medica, Bologna, Emilia-Romagna
  - Ospedale Bufalini, Forlì, Emilia-Romagna
  - Fondazione IRCCS Istituto Neurologico C. Besta; Neuro-oncologia Sperimentale e Terapia Genica, Milan, Lombardy
  - Azienda Ospedaliera Le Molintte di Torino; Dipartimento Di Neurologia - Oncologia, Turin, Piedmont
  - Az. Osp. S. Maria; Dept. Di Oncologia Medica, Terni, Umbria
  - Ospedale di Treviso, Universita di Padova; Neurosurgery Dept, Treviso, Veneto
- Japan (8):
  - Hiroshima University Hospital; Neurosurgery, Hiroshima
  - Tsukuba University Hospital; Neurology, Ibaraki
  - Kumamoto University Hospital; Neurosurgery, Kumamoto
  - Kitano Hospital; Neurosurgery, Osaka
  - Saitama Medical University International Medical Center; Clinical and Medical Oncology, Saitama
  - National Cancer Center Hospital; Neurosurgery, Tokyo
  - Komagome Hospital; Neurosurgery, Tokyo
  - Kyorin University Hospital; Neurosurgery, Tokyo
- Netherlands (3):
  - VU MEDISCH CENTRUM; Dept. of Medical Oncology, Amsterdam
  - Catharina Ziekenhuis; Dept of Internal Medicin, Eindhoven
  - Utrecht University Medical Centre; Dept of Medical Oncology and UPC, Utrecht
- New Zealand (3):
  - Auckland city hospital; Auckland Regional Cancer Centre and Blood Service, Auckland
  - Christchurch Hospital; Dept of Oncology, Christchurch
  - Waikato Hospital; Regional Cancer Center, Hamilton
- Poland (3):
  - Bialostockie Centrum Onkologii; Oddzial Onkologii Klinicznej, Bialystok
  - Centrum Onkologii;Im. Franciszka Lukaszczyka;Onkologii, Bydgoszcz
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie; Klinika Neurochirurgii i Neurochirurgii Dzi, Lublin
- Portugal (4):
  - IPO de Coimbra; Servico de Oncologia Medica, Coimbra
  - IPO de Lisboa; Servico de Neurologia, Lisbon
  - Hospital de Santa Maria; Servico de Oncologia Medica, Lisbon
  - Hospital de Sao Joao; Servico de Oncologia, Porto
- Romania (3):
  - Institut Oncologic Prof. Dr. Alexandru Trestioreanu; Departament Radioterapie, Bucharest
  - Institut Oncologic Ion Chiricuta; Departament Radioterapie, Cluj-Napoca
  - Spital Clinic Judetean Mures; Oncologie, Târgu Mureş
- Russia (4):
  - N.N.Burdenko Main Military Clinical Hospital; Oncology Dept, Moscow
  - Russian Research Oncology Center n.a. N.N. Blokhin of the RAMS; Department of Neurosurgery, Moscow
  - Scientific Research Neurosurgery Institute; Dept. of Neurooncology, Moscow
  - Institution of Higher Professional Learning Military; Neurooncology, Saint Petersburg
- South Korea (8):
  - Pusan National University Hospital; Neuro Sugery, Busan
  - Kyungpook National University Hosital; Neuro Sugery, Daegu
  - National Cancer Centre; Neurosurgery Dept, Goyang-si
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National Uni Hospital; Dept. of Internal Medicine/Hematology/Oncology, Seoul
  - Asan Medical Center; Medical Oncology, Seoul
  - Yonsei University Severance Hospital; Medical Oncology, Seoul
  - Samsung Medical Center; Neurosurgery Department, Seoul
- Spain (7):
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Barcelona
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Regional Universitario Carlos Haya; Servicio de Oncologia, Málaga
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
- Sweden (4):
  - Sahlgrenska Universitetssjukhuset; Jubileumskliniken, Gothenburg
  - Skånes University Hospital, Skånes Department of Onclology, Lund
  - Norrlands Universitetssjukhus; Cancer Centrum, Umeå
  - Akademiska sjukhuset, Onkologkliniken, Uppsala
- HUG; Oncologie, Geneva, Switzerland
- United Kingdom (9):
  - Queen Elizabeth Medical Centre; Neurosurgery, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - The Royal Marsden NHS Foundation Trust; Oncology, London
  - The Clatterbridge Cancer Ctr For Oncolgy, Metropolitan Borough of Wirral
  - Northern Centre for Cancer Care;Oncology, Newcastle upon Tyne
  - Nottingham City Hospital; Dept of Haematology, Nottingham
  - Queen's Hospital; Oncology, Romford
  - Weston Park Hospital; Cancer Clinical Trials Centre, Sheffield
  - Royal Marsden Hospital; Dept of Medical Oncology, Sutton

REFERENCES:
- [Derived] Seliger C, Oppong FB, Lefranc F, Chinot O, Stupp R, Nabors B, Gorlia T, Weller M; EORTC Brain Tumor Group. Association of antidepressant drug use with outcome of patients with glioblastoma. Int J Cancer. 2023 Apr 1;152(7):1348-1359. doi: 10.1002/ijc.34344. Epub 2022 Nov 17. PMID 36346112
- [Derived] Hagiwara A, Schlossman J, Shabani S, Raymond C, Tatekawa H, Abrey LE, Garcia J, Chinot O, Saran F, Nishikawa R, Henriksson R, Mason WP, Wick W, Cloughesy TF, Ellingson BM. Incidence, molecular characteristics, and imaging features of "clinically-defined pseudoprogression" in newly diagnosed glioblastoma treated with chemoradiation. J Neurooncol. 2022 Sep;159(3):509-518. doi: 10.1007/s11060-022-04088-3. Epub 2022 Jul 17. PMID 35842871
- [Derived] Jiguet-Jiglaire C, Boissonneau S, Denicolai E, Hein V, Lasseur R, Garcia J, Romain S, Appay R, Graillon T, Mason W, Carpentier AF, Brandes AA, Ouafik L', Wick W, Baaziz A, Gigan JP, Arguello RJ, Figarella-Branger D, Chinot O, Tabouret E. Plasmatic MMP9 released from tumor-infiltrating neutrophils is predictive for bevacizumab efficacy in glioblastoma patients: an AVAglio ancillary study. Acta Neuropathol Commun. 2022 Jan 3;10(1):1. doi: 10.1186/s40478-021-01305-4. PMID 34980260
- [Derived] Chinot OL, Nishikawa R, Mason W, Henriksson R, Saran F, Cloughesy T, Garcia J, Revil C, Abrey L, Wick W. Upfront bevacizumab may extend survival for glioblastoma patients who do not receive second-line therapy: an exploratory analysis of AVAglio. Neuro Oncol. 2016 Sep;18(9):1313-8. doi: 10.1093/neuonc/now046. Epub 2016 Mar 22. PMID 27006178
- [Derived] Saran F, Chinot OL, Henriksson R, Mason W, Wick W, Cloughesy T, Dhar S, Pozzi E, Garcia J, Nishikawa R. Bevacizumab, temozolomide, and radiotherapy for newly diagnosed glioblastoma: comprehensive safety results during and after first-line therapy. Neuro Oncol. 2016 Jul;18(7):991-1001. doi: 10.1093/neuonc/nov300. Epub 2016 Jan 24. PMID 26809751
- [Derived] Taphoorn MJ, Henriksson R, Bottomley A, Cloughesy T, Wick W, Mason WP, Saran F, Nishikawa R, Hilton M, Theodore-Oklota C, Ravelo A, Chinot OL. Health-Related Quality of Life in a Randomized Phase III Study of Bevacizumab, Temozolomide, and Radiotherapy in Newly Diagnosed Glioblastoma. J Clin Oncol. 2015 Jul 1;33(19):2166-75. doi: 10.1200/JCO.2014.60.3217. Epub 2015 May 26. PMID 26014298
- [Derived] Chinot OL, Wick W, Mason W, Henriksson R, Saran F, Nishikawa R, Carpentier AF, Hoang-Xuan K, Kavan P, Cernea D, Brandes AA, Hilton M, Abrey L, Cloughesy T. Bevacizumab plus radiotherapy-temozolomide for newly diagnosed glioblastoma. N Engl J Med. 2014 Feb 20;370(8):709-22. doi: 10.1056/NEJMoa1308345. PMID 24552318
- [Derived] Chinot OL, Macdonald DR, Abrey LE, Zahlmann G, Kerloeguen Y, Cloughesy TF. Response assessment criteria for glioblastoma: practical adaptation and implementation in clinical trials of antiangiogenic therapy. Curr Neurol Neurosci Rep. 2013 May;13(5):347. doi: 10.1007/s11910-013-0347-2. PMID 23529375

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The primary completion date for co-primary outcome of Progression-Free Survival (PFS) was 31 Mar 2012, whereas, the primary completion date for co-primary outcome of Overall Survival (OS) was 28 Feb 2013. Data for PFS and OS are reported according to these cut-off dates.
Groups:
- Bevacizumab + RT + Temozolomide: In the Concurrent Phase participants received radiotherapy (RT) in daily fractions of 2 Gray (Gy) given 5 days per weeks for 6 weeks (for a total of 60 Gy) and temozolomide 75 milligrams per square meter (mg/m^2) daily from the first day to the last day of radiotherapy (for a maximum of 49 days in case of delay to the end of radiation therapy) and bevacizumab (Avastin) 10 milligrams per kilogram (mg/kg) intravenous (IV) every 2 weeks for 6 weeks. There was a 4 week treatment break. Participants then entered the Maintenance Phase where they received six 28-day cycle of bevacizumab 10 mg/kg IV every 2 weeks and temozolomide 150 to 200 mg/m^2 daily in the first 5 days of each cycle. The participants then entered the Monotherapy Phase where they received bevacizumab 15 mg/kg IV every 3 weeks until disease progression/unacceptable toxicity. Participants then entered the last period: After Primary Overall Survival Analysis, in which participants were followed up for safety.
- Placebo + RT + Temozolomide: In the Concurrent Phase participants received radiotherapy in daily fractions of 2 Gy given 5 days per week for 6 weeks (for a total of 60 Gy) and temozolomide 75 mg/m^2 daily from the first day to the last day of radiotherapy (for a maximum of 49 days in case of delay to the end of radiation therapy) and placebo IV every 2 weeks for 6 weeks. There was a 4 week treatment break. Participants then entered the Maintenance Phase where they received six 28-day cycle of placebo IV every 2 weeks and temozolomide 150 to 200 mg/m^2 daily in the first 5 days of each cycle. The participants then entered the Monotherapy Phase where they received placebo IV every 3 weeks until disease progression/unacceptable toxicity. Participants then entered the last period: After Primary Overall Survival Analysis, in which participants were followed up for safety.
Period: Concurrent Phase
Arm/Group | Bevacizumab + RT + Temozolomide | Placebo + RT + Temozolomide
Started | 458 | 463
Treated | 452 | 459
Completed | 397 | 421
Not Completed | 61 | 42
Not completed — Adverse Event | 50 | 27
Not completed — Withdrew consent | 3 | 7
Not completed — Refused treatment/Did not cooperate | 5 | 7
Not completed — Administrative reasons | 2 | 1
Not completed — Protocol Violation | 1 | 0
Period: Maintenance Phase
Arm/Group | Bevacizumab + RT + Temozolomide | Placebo + RT + Temozolomide
Started | 396 (Some who completed previous period had discontinued, progressed, or died prior to this period.) | 370 (Some who completed previous period had discontinued, progressed, or died prior to this period.)
Completed | 353 | 331
Not Completed | 43 | 39
Not completed — Adverse Event | 31 | 30
Not completed — Withdrew consent | 2 | 4
Not completed — Refused treatment/Did not cooperate | 6 | 3
Not completed — Administrative reasons | 4 | 1
Not completed — Failure to return | 0 | 1
Period: Monotherapy Phase
Arm/Group | Bevacizumab + RT + Temozolomide | Placebo + RT + Temozolomide
Started | 269 (Some who completed previous period had discontinued, progressed, or died prior to this period.) | 159 (Some who completed previous period had discontinued, progressed, or died prior to this period.)
Completed | 204 | 143
Not Completed | 65 | 16
Not completed — Adverse Event | 42 | 5
Not completed — Administrative reasons | 11 | 5
Not completed — Refused treatment/ Did not cooperate | 8 | 2
Not completed — Withdrew Consent | 2 | 3
Not completed — Failure to return | 2 | 1
Period: After Primary Overall Survival Analysis
Arm/Group | Bevacizumab + RT + Temozolomide | Placebo + RT + Temozolomide
Started | 27 (Some who completed previous period had discontinued, progressed, or died prior to this period.) | 20 (Some who completed previous period had discontinued, progressed, or died prior to this period.)
Completed | 0 | 0
Not Completed | 27 | 20
Not completed — Adverse Event | 11 | 0
Not completed — Administrative reasons | 10 | 16
Not completed — Progression of Disease | 2 | 4
Not completed — Withdrew Consent | 4 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population included all randomized participants.
Groups:
- Placebo + RT +Temozolomide: In the Concurrent Phase participants received RT in daily fractions of 2 Gy given 5 days per weeks for 6 weeks (for a total of 60 Gy) and temozolomide 75 mg/m^2 daily from the first day to the last day of radiotherapy (for a maximum of 49 days in case of delay to the end of radiation therapy) and placebo IV every 2 weeks for 6 weeks. There was a 4 week treatment break. Participants then entered the Maintenance Phase where they received six 28-day cycle of placebo IV every 2 weeks and temozolomide 150 to 200 mg/m^2 daily in the first 5 days of each cycle. The participants then entered the Monotherapy Phase where they received placebo IV every 3 weeks until disease progression/unacceptable toxicity. Participants then entered the last period: After Primary Overall Survival Analysis, in which participants were followed up for safety.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + RT + Temozolomide | Placebo + RT +Temozolomide | Total
Number analyzed (Participants) | 458 | 463 | 921
Age, Continuous [Mean (Full Range); unit: years] | 55.9 [20 to 84] | 55.9 [18 to 79] | 55.9 [18 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 165 | 341
  Male | 282 | 298 | 580

OUTCOME MEASURES:

1. Primary Outcome: Co-Primary: Progression-free Survival (PFS) as Assessed by Investigator
Description: PFS is defined as time from randomization to disease progression (PD) or death. PD was assessed using adapted Macdonald response criteria (modified World Health Organization [WHO] criteria) based on 3 components: radiological tumor assessments using Magnetic Resonance Imaging [MRI] scans,neurological assessment and changes in corticosteroid use. PD is assessed as greater than or equal to(>=) 25% increase in sum of products of the longest diameters of all index lesions (enhancing,measurable) compared with the smallest recorded sum (nadir); or unequivocal PD of existing non-index lesions (non-enhancing and enhancing,non-measurable); or unequivocal appearance of new lesions); or neurological worsening (if corticosteroid dose is stable or increased) compared to neurological evaluation at previous disease assessment with no need for a confirmatory scan. Participants without a PFS event were censored at last disease assessment.
Time Frame: Randomization until PFS Event [Until data cutoff= 31 March 2012 (up to 31.4 months)
Population: Intent to treat population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + RT + Temozolomide | Placebo + RT + Temozolomide
Number analyzed (Participants) | 458 | 463
Months | 10.6 [10.0 to 11.4] | 6.2 [6.0 to 7.5]
Statistical Analysis 1: Comparison: Bevacizumab + RT + Temozolomide vs Placebo + RT + Temozolomide; Test type: Superiority or Other; p < 0.0001, Log Rank — Stratified by Region and Recursive partitioning analysis (RPA) Class; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.55 to 0.74] — Stratified by Region and RPA Class

2. Primary Outcome: Co-Primary: Overall Survival (OS)
Description: Overall Survival was defined as the time from randomization to death due to any cause.
Time Frame: Randomization until OS Event (Until data cutoff= 28 February 2013 [up to 42.2 months])
Population: Intent to treat population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + RT + Temozolomide | Placebo + RT + Temozolomide
Number analyzed (Participants) | 458 | 463
Months | 16.8 [15.5 to 18.5] | 16.7 [15.4 to 18.4]
Statistical Analysis 1: Comparison: Bevacizumab + RT + Temozolomide vs Placebo + RT + Temozolomide; Test type: Superiority or Other; p = 0.0987, Log Rank; Stratified by Region and RPA Class; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.76 to 1.02] — Stratified by Region and RPA Class

3. Secondary Outcome: PFS as Assessed by an Independent Review Facility
Description: An Independent Review Facility reviewed the MRI scans used by investigator to evaluate radiological tumor response. PFS is defined as time from randomization to PD or death. PD was assessed using adapted Macdonald response (modified WHO) criteria based on 3 components: radiological tumor assessments using MRI scans, neurological assessment and changes in corticosteroid use. PD is assessed as >=25% increase in sum of products of the longest diameters of all index lesions (enhancing, measurable) compared with the smallest recorded sum (nadir); or unequivocal PD of existing non-index lesions (non-enhancing and enhancing, non-measurable); or unequivocal appearance of new lesions); or neurological worsening (if corticosteroid dose is stable or increased) compared to neurological evaluation at previous disease assessment with no need for a confirmatory scan. Participants without a PFS event were censored at last disease assessment.
Time Frame: Randomization until PFS Event (Until data cutoff= 31 March 2012 [up to 29.5 months])
Population: Intent to treat population.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Bevacizumab + RT +Temozolomide: In the Concurrent Phase participants received RT in daily fractions of 2 Gy given 5 days per weeks for 6 weeks (for a total of 60 Gy) and temozolomide 75 mg/m^2 daily from the first day to the last day of radiotherapy (for a maximum of 49 days in case of delay to the end of radiation therapy) and bevacizumab 10 mg/kg IV every 2 weeks for 6 weeks. There was a 4 week treatment break. Participants then entered the Maintenance Phase where they received six 28-day cycle of bevacizumab 10 mg/kg IV every 2 weeks and temozolomide 150 to 200 mg/m^2 daily in the first 5 days of each cycle. The participants then entered the Monotherapy Phase where they received bevacizumab 15 mg/kg IV every 3 weeks until disease progression/unacceptable toxicity.
Arm/Group | Bevacizumab + RT +Temozolomide | Placebo + RT + Temozolomide
Number analyzed (Participants) | 458 | 463
Months | 8.4 [7.9 to 9.7] | 4.3 [4.1 to 5.1]
Statistical Analysis 1: Comparison: Bevacizumab + RT +Temozolomide vs Placebo + RT + Temozolomide; Test type: Superiority or Other; p < 0.0001, Log Rank — Stratified by Region and RPA Class; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.53 to 0.71] — Stratified by Region and RPA Class

4. Secondary Outcome: Kaplan-Meier (KM) Estimate of One Year Overall Survival
Description: KM estimate of one year overall survival (probability to survive for at least 1 year) was reported. Corresponding 95% confidence interval (CI) was calculated using Greenwood's formula.
Time Frame: Randomization until Overall Survival Event (Until data cutoff= 28 February 2013 [up to 42.2 months])
Population: Intent to treat population.
Measure: Number (95% Confidence Interval); unit: probability of being alive
Arm/Group | Bevacizumab + RT + Temozolomide | Placebo + RT + Temozolomide
Number analyzed (Participants) | 458 | 463
probability of being alive | 0.72 [0.68 to 0.77] | 0.66 [0.62 to 0.71]

5. Secondary Outcome: Kaplan-Meier (KM) Estimate of Two Year Overall Survival
Description: KM estimate of two year overall survival was reported (probability to survive for at least 2 years). Corresponding 95% CI was calculated using Greenwood's formula.
Time Frame: Randomization until Overall Survival Event (Until data cutoff= 28 February 2013 [up to 42.2 months])
Population: Intent to treat population.
Measure: Number (95% Confidence Interval); unit: probability of being alive
Arm/Group | Bevacizumab + RT + Temozolomide | Placebo + RT + Temozolomide
Number analyzed (Participants) | 458 | 463
probability of being alive | 0.34 [0.29 to 0.38] | 0.30 [0.26 to 0.34]

6. Secondary Outcome: PFS in Participants With Stable/Improved Health Related Quality of Life (HRQoL) Based on European Organization for Research & Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core 30 (C30)(EORTC QLQ-C30) & EORTC QLQ Brain Neoplasm 20 (BN20)
Description: EORTC QLQ-C30: 30 items; 5 functional scales; 9 symptom scales; & global health status. Most questions used 4-point scale (1:Not at all, 4:Very much), 2 questions used 7-point scale (1:very poor, 7:Excellent). EORTC QLQ-BN20: 20 items rated on a 4 point scale (1:not at all, 4:very much). EORTC QLQ-C30 and BN20 scores were transformed to a 0-100 scale, higher score=better functioning/global health (C30) or more severe symptoms (BN20). Stable HRQoL: change from baseline (BL) within 10 points. Improved HRQoL: an increase from BL >/=10 points for functioning/global health status, & decrease of >/=10 points for symptoms. PFS is reported for participants with Stable/Improved global health; physical, social functioning (C30); motor dysfunction & communication deficit (BN20). PFS: randomization to PD or death. PD: >=25% increase in sum of products of longest diameters of index lesions; or progression of existing non-index lesions; or appearance of new lesions; or neurological worsening.
Time Frame: Randomization until PFS Event [Until data cutoff= 31 March 2012 (up to 31.4 months)
Population: Intent to treat population. Number of Participants Analyzed = overall participants evaluable for this outcome measure; n = participants evaluable for specified category.
Measure: Median (Full Range); unit: Months
Arm/Group | Bevacizumab + RT + Temozolomide | Placebo + RT + Temozolomide
Number analyzed (Participants) | 458 | 463
Months
  Global health status (n=354, 309) | 8 [0 to 26] | 4 [1 to 29]
  Physical functioning (n=353, 318) | 7 [0 to 27] | 5 [1 to 29]
  Social functioning (n=352, 327) | 8 [0 to 26] | 4 [0 to 27]
  Motor dysfunction (n=361, 314) | 7 [1 to 27] | 4 [0 to 26]
  Communication deficit (n=365, 329) | 8 [0 to 27] | 4 [1 to 24]

7. Secondary Outcome: Number of Participants With Non-Serious Adverse Events, Serious Adverse Events and Death
Description: An adverse event (AE) was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as AE.A serious adverse event (SAE) is any experience that suggests a significant hazard,contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant. Non-serious adverse events (Non-SAEs) included all AEs except SAEs (non-SAEs = all AEs - SAEs). Nine participants randomized to the Placebo+RT+Temozolomide arm incorrectly received at least 1 dose of bevacizumab and were added to the Bevacizumab+RT+Temozolomide arm for Safety.
Time Frame: Randomization until study completion (Until data cutoff= 09 Sep 2015 [up to 64 months])
Population: Safety Population included all randomized participants who received study treatment during the treatment period (10 participants did not receive at least one dose of study treatment and were therefore excluded, 4 in Placebo and 6 in Bevacizumab.
Measure: Number; unit: Participants
Arm/Group | Bevacizumab + RT + Temozolomide | Placebo + RT + Temozolomide
Number analyzed (Participants) | 461 | 450
Participants
  Non-SAEs | 437 | 412
  SAEs | 179 | 115
  Death | 335 | 337

ADVERSE EVENTS:
Time Frame: Randomization until study completion (Until data cutoff= 09 Sep 2015 [up to 64 months])
Description: Safety Population.10 participants did not receive at least 1 dose of drug and were excluded, 4 in Placebo and 6 in Bevacizumab.9 participants randomized to the Placebo+RT+Temozolomide arm incorrectly received at least 1 dose of bevacizumab and were added to the Bevacizumab+RT+Temozolomide arm for safety.Other AEs are non-SAEs (AEs excluding SAEs).
Groups:
- Bevacizumab + RT+Temozolomide: In the Concurrent Phase participants received radiotherapy in daily fractions of 2 Gy given 5 days per weeks for 6 weeks (for a total of 60 Gy) and temozolomide 75 mg/m^2 daily from the first day to the last day of radiotherapy (for a maximum of 49 days in case of delay to the end of radiation therapy) and bevacizumab 10 mg/kg intravenous (IV) every 2 weeks for 6 weeks. There was a 4 week treatment break. Participants then entered the Maintenance Phase where they received six 28-day cycle of bevacizumab 10 mg/kg IV every 2 weeks and temozolomide 150 to 200 mg/m^2 daily in the first 5 days of each cycle. The participants then entered the Monotherapy Phase where they received bevacizumab 15 mg/kg IV every 3 weeks until disease progression/unacceptable toxicity. Participants then entered the last period: After Primary Overall Survival Analysis, in which participants were followed up for safety.
- Placebo + RT+Temozolomide: In the Concurrent Phase participants received radiotherapy in daily fractions of 2 Gy given 5 days per weeks for 6 weeks (for a total of 60 Gy) and temozolomide 75 mg/m^2 daily from the first day to the last day of radiotherapy (for a maximum of 49 days in case of delay to the end of radiation therapy) and placebo IV every 2 weeks for 6 weeks. There was a 4 week treatment break. Participants then entered the Maintenance Phase where they received six 28-day cycle of placebo IV every 2 weeks and temozolomide 150 to 200 mg/m^2 daily in the first 5 days of each cycle. The participants then entered the Monotherapy Phase where they received placebo IV every 3 weeks until disease progression/unacceptable toxicity. Participants then entered the last period: After Primary Overall Survival Analysis, in which participants were followed up for safety.
Arm/Group | Bevacizumab + RT+Temozolomide | Placebo + RT+Temozolomide
Serious Adverse Events (participants affected / at risk) | 179/461 | 115/450
Other Adverse Events (participants affected / at risk) | 437/461 | 412/450
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + RT+Temozolomide (N=461) | Placebo + RT+Temozolomide (N=450)
Pneumonia (Infections and infestations) | 10 | 5
Sepsis (Infections and infestations) | 6 | 1
Urinary tract infection (Infections and infestations) | 1 | 3
Brain abscess (Infections and infestations) | 1 | 3
Lower respiratory tract infection (Infections and infestations) | 0 | 3
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 2
Postoperative wound infection (Infections and infestations) | 3 | 0
Respiratory tract infection (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 2 | 1
Infection (Infections and infestations) | 2 | 0
Meningitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 3 | 0
Abscess (Infections and infestations) | 1 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Encephalitis herpes (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Graft infection (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oral fungal infection (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Convulsion (Nervous system disorders) | 5 | 6
Cerebrovascular accident (Nervous system disorders) | 8 | 2
Brain oedema (Nervous system disorders) | 2 | 4
Headache (Nervous system disorders) | 4 | 2
Cerebral ischaemia (Nervous system disorders) | 3 | 2
Epilepsy (Nervous system disorders) | 3 | 2
Ischaemic stroke (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 2
Hemiparesis (Nervous system disorders) | 1 | 1
Hydrocephalus (Nervous system disorders) | 2 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 1
Neurological decompensation (Nervous system disorders) | 1 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Basal ganglia stroke (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral thrombosis (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 8
Neutropenia (Blood and lymphatic system disorders) | 4 | 2
Pancytopenia (Blood and lymphatic system disorders) | 5 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 2
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 13 | 12
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Anal prolapse (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Rectal perforation (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 11 | 6
Hypertension (Vascular disorders) | 4 | 1
Venous thrombosis (Vascular disorders) | 0 | 2
Embolism (Vascular disorders) | 1 | 0
Embolism venous (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 2 | 0
Thrombosis (Vascular disorders) | 1 | 0
Pyrexia (General disorders) | 8 | 3
General physical health deterioration (General disorders) | 3 | 2
Fatigue (General disorders) | 0 | 2
Cyst (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 5
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Acute psychosis (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Delirium tremens (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Diabetes insipidus (Endocrine disorders) | 0 | 1
Troponin increased (Investigations) | 0 | 1
Scrotal cyst (Reproductive system and breast disorders) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Optic Neuropathy (Eye disorders) | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Extradural Abscess (Infections and infestations) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + RT+Temozolomide (N=461) | Placebo + RT+Temozolomide (N=450)
Nausea (Gastrointestinal disorders) | 223 | 191
Constipation (Gastrointestinal disorders) | 178 | 137
Vomiting (Gastrointestinal disorders) | 145 | 100
Diarrhoea (Gastrointestinal disorders) | 95 | 69
Abdominal pain (Gastrointestinal disorders) | 33 | 17
Dyspepsia (Gastrointestinal disorders) | 31 | 16
Abdominal pain upper (Gastrointestinal disorders) | 35 | 12
Gingival bleeding (Gastrointestinal disorders) | 36 | 6
Fatigue (General disorders) | 191 | 178
Asthenia (General disorders) | 86 | 63
Oedema peripheral (General disorders) | 36 | 34
Pyrexia (General disorders) | 39 | 26
Alopecia (Skin and subcutaneous tissue disorders) | 180 | 162
Rash (Skin and subcutaneous tissue disorders) | 76 | 60
Pruritus (Skin and subcutaneous tissue disorders) | 54 | 37
Dry skin (Skin and subcutaneous tissue disorders) | 34 | 24
Headache (Nervous system disorders) | 172 | 130
Dizziness (Nervous system disorders) | 46 | 53
Dysgeusia (Nervous system disorders) | 39 | 33
Convulsion (Nervous system disorders) | 36 | 39
Thrombocytopenia (Blood and lymphatic system disorders) | 148 | 120
Neutropenia (Blood and lymphatic system disorders) | 66 | 53
Leukopenia (Blood and lymphatic system disorders) | 56 | 40
Lymphopenia (Blood and lymphatic system disorders) | 34 | 39
Anaemia (Blood and lymphatic system disorders) | 27 | 34
Arthralgia (Musculoskeletal and connective tissue disorders) | 71 | 30
Pain in extremity (Musculoskeletal and connective tissue disorders) | 48 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 29
Muscular weakness (Musculoskeletal and connective tissue disorders) | 29 | 33
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 39 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 98 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 55 | 46
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 42 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 29 | 12
Hypertension (Vascular disorders) | 175 | 51
Decreased appetite (Metabolism and nutrition disorders) | 116 | 74
Insomnia (Psychiatric disorders) | 53 | 42
Depression (Psychiatric disorders) | 43 | 30
Anxiety (Psychiatric disorders) | 29 | 25
Nasopharyngitis (Infections and infestations) | 63 | 26
Urinary tract infection (Infections and infestations) | 49 | 27
Upper respiratory tract infection (Infections and infestations) | 31 | 13
Weight decreased (Investigations) | 36 | 18
Alanine aminotransferase increased (Investigations) | 22 | 25
Proteinuria (Renal and urinary disorders) | 72 | 19
Radiation skin injury (Injury, poisoning and procedural complications) | 38 | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.